CLINICAL TRIAL: NCT01598779
Title: Human Papillomavirus (HPV) Types Present in External Genital Warts (EGW) in the Argentinean Population
Status: Completed | Type: Observational
Sponsor: University of Buenos Aires (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Laura Alicia Fleider, Physician, University of Buenos Aires
Other Study IDs: Genital Warts
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Condylomata Acuminata
Keywords: genital warts; HPV types; Sexually Transmitted Diseases; Skin Diseases, Viral; Tumor Virus Infections; Skin Diseases, Infectious; Skin Diseases; Papillomavirus Infections; DNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral
MeSH Terms: conditions — Condylomata Acuminata; Sexually Transmitted Diseases; Skin Diseases, Viral; Tumor Virus Infections; Skin Diseases, Infectious; Skin Diseases; Papillomavirus Infections; DNA Virus Infections; Virus Diseases; Sexually Transmitted Diseases, Viral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy specimens will be held in a formol 10% solution and will be sent to the pathologist. A portion of each sample will be processed for histological analysis, which will be performed by one pathologist. The remainder of each specimen will be saved to extract DNA for PCR analysis
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The summary of this study is to know which HPV types are present in genital warts in Argentinean population.

DETAILED DESCRIPTION:
This is a prospective study. Patients will be evaluated for the presence of external anogenital warts in our clinic. Biopsy will be performed if patients have genital lesions consistent with genital warts of the external genitalia or perianal area. All patients will be provided with an informed consent for the excision biopsy procedure, before performing the biopsy of the lesion. Biopsy specimens will be held in a formol 10% solution and will be sent to the pathologist. A portion of each sample will be processed for histological analysis, which will be performed by one pathologist. The remainder of each specimen will be saved to extract DNA for PCR analysis. All biopsies will be analyzed by the same pathologist who will confirm the histology of the lesion. A part of the specimen will be kept frozen and if the biopsy confirm genital warts by histology; then the specimen will be analyzed by PCR for the presence of DNA HPV 6 and 11. The PCR analysis will be done by microarrays. Detection is performed in a subtype of array platform system which detects the different types of virus. The reports will be as undetectable / detectable and type.

The study will be conducted in the Institute of Gynecology and Fertility (Institute affiliated with the School of Medicine - University of Buenos Aires).

Chronogram of activities: all activities will be done in a maximum of 60 days

1. st visit: detect external genital warts and firm informed consent and take the biopsy
2. nd visit: inform the result

ELIGIBILITY:
Inclusion Criteria:

* women between 15 and 45 years old, with External Genital Warts

Exclusion Criteria:

* women taking corticoid therapy, having an immunosuppressed disease, pregnancy, cancer related to HPV, VIN confirmed by histology, other sexually transmitted infection, HIV+ known

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Women with genital warts
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Fleider, MD, Principal Investigator — University of Buenos Aires; Laura A Fleider, MD, Principal Investigator — Institute of Gynecology and Fertility
Locations (1):
- IFER, Buenos Aires, Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Having External Genital Warts: Patients were examined by experienced ginecologists in their first visit to evaluate the presence of lesions suspicious of condilomata acuminate, If they had lesions suspicious of gential warts, they were invited to participate and given an informed consent. Biopsied from genital warts were taken with an excisional procedure under local anesthesia. Biopsied sample was splinted in order to obtain two pieces, one of them was kept in formol solution (10%) and sent to the pathology laboratory for hematoxiline - eosine paint and lecture. All biopsies were analyzed by expert pathologists in order to confirm the histological diagnosis of genital warts. The other piece was sent to the laboratory to investigate the presence of HPV 6 and 11.
  In this first visit, the chronogram of activities included the detection of external genital warts, review of the criteria for inclusion and exclusion, firm informed consent, complete the questionnaire and take the biopsy, on a 2nd visit we informed the
Period: Overall Study
Arm/Group | Patients Having External Genital Warts
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Women age 15-45 attending an outpatient consultation at clinics of the investigators or at University of Buenos Aires, with a lesion suspected of being HPV related.
Arm/Group | Patients Having External Genital Warts
Number analyzed (Participants) | 150
Age, Continuous [Mean (Full Range); unit: years] — Women age 15-45 years, with a lesion suspected of being HPV related were eligible to enter in the study.
  years | 28.48 [15 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 150

OUTCOME MEASURES:

1. Primary Outcome: Human Papillomavirus (HPV) Types in External Genital Warts (EGW)
Description: 150 biopsies with histological diagnosis of genital warts were analyzed by PCR to detect HPV type
Time Frame: 4 months
Population: Biopsied from genital warts were taken with an excisional procedure under local anesthesia. Biopsied sample was splinted in order to obtain two pieces, All biopsies were analyzed to confirm the histological diagnosis of genital warts. The other piece was sent to the laboratory to investigate the presence of HPV 6 and 11.
Measure: Number; unit: percentage of participants
Groups:
- Women With External Genital Warts: Women age 15-45 attending an outpatient consultation at clinics of the investigators or at University of Buenos Aires, with a lesion suspected of being HPV related were eligible to enter in the study. The main manifestations of genital warts include cauliflower-like condylomata acuminata lesions, keratotic and smooth papular warts, subclinical "flat" warts, Patients previously vaccinated with commercially available vaccines (Gardasil™ or Cervarix™) were not invited to participate.
  Inclusion criteria: women between 15 and 45 years old, with External Genital Warts. We will exclude women under treatment corticosteroids, having an immunosuppressive disease, pregnancy, cancer related to HPV, VIN confirmed by histology, other sexually transmitted infection, HIV+ known
Arm/Group | Women With External Genital Warts
Number analyzed (Participants) | 150
percentage of participants
  HPV 6 | 80
  HPV 11 | 12.66
  HPV 6 & 11 | 0.66
  HPV 16 | 2
  HPV 73 | 0.66
  Negative | 4

ADVERSE EVENTS:
Arm/Group | Patients Having External Genital Warts
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 0/150

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No